CLINICAL TRIAL: NCT02235766
Title: Corelab Remotely Echocardiographic Imaging Acquisition in Cardiac Resynchronization Therapy Candidates
Acronym: CORELAB-CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kell s.r.l. (Other)
Responsible Party: Sponsor
Other Study IDs: Kell-1
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Satellite Tele-Echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT candidates patients: In accordance with the current ESC/ACCF/AHA indications for CRT in sinus rhythm, all patients in NYHA class II, III and IV with QRS complex greater than 120 msec and ejection fraction equal or less than 35% will be considered eligible to participate in this observational study.
  Interventions: Other: Echocardiographic assessment

INTERVENTIONS:
Other: Echocardiographic assessment

SUMMARY:
Purpose of the observational study is to assess the capability of a satellite tele-echocardiography (STE) system to acquire and transmit echocardiographic images and clips to an echocardiographic core laboratory (ECL) in a real time mode without loss of quality. Additionally the prognostic efficacy of specific echo parameters in the cardiac resynchronization therapy response will be evaluated.

DETAILED DESCRIPTION:
CORELAB-CRT is a prospective multi center Italian observational study. All echo images and clips will be transmitted by using an integrated satellite transmission system. All echo assessments performed in accordance to the centers clinical practice will be also used to investigate the prognostic efficacy of echo parameters in term of response to the cardiac resynchronization therapy (CRT). All commercially available multi-chamber CRT-D devices from any manufacturers are allowed in this observational study.

Any compatible market released right atrial, right ventricular and left ventricular lead from any manufacturer is allowed.

The echocardiography device models used to perform echo imaging for all patients participating in this analysis are GE Vivid 7, GE Vivid 9 and GE Vivid I, according to the model used in the clinical practice of the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA class II, III and ambulatory IV with:

   * QRS complex duration ≥120msec;
   * Ejection fraction ≤35%.
2. Optimized medical treatment;
3. Patient in sinus rhythm;
4. Patient is willing and able to sign an informed consent form.

Exclusion Criteria:

1. Unstable angina, or acute myocardial infarction, coronary-aortic bypass graft or percutaneous transluminal coronary angioplasty within the past 3 months;
2. Cerebral vascular attacks or transient ischemic attack within the last month;
3. Chronic atrial arrhythmias, paroxysmal atrial fibrillation events;
4. Patients already implanted with an ICD or a CRT device;
5. Pacemaker dependency or ventricular pacing percentage ≥10%;
6. Valvular disease with an indication for surgical correction ≤12 months survival expectancy;
7. Mechanical right ventricular valve;
8. Patient is enrolled in or intends to participate in another clinical trial that may have an impact on the study endpoints;
9. Pregnancy or breastfeeding;
10. Previous heart transplant;
11. Refusal of study informed consent;
12. Expected lack of compliance during follow-up;
13. Patient is less than 18 years of age;
14. Patient's life expectancy is less than 6 months in the opinion of physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In accordance with the current ESC/ACCF/AHA indications for CRT in sinus rhythm, all patients in NYHA class II, III and IV with QRS complex greater than 120 msec and ejection fraction equal or less than 35% will be considered eligible to participate in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
ECM assessment | 6 months
  Agreement in the echocardiographic measurement capability (EMC) between transmitted and echocardiographic device image on the set of high quality images transmitted by STE. Each echo image will be classified as high quality image if the Mean Opinion Score (MOS) will be greater than 3 points. For each high quality echo image (MOS greater or equal 3) the EMC will be assessed to both transmitted and device echocardiographic image.

SECONDARY OUTCOMES:
Prognostic efficacy of specific echo parameters | 6 months
  Echocardiographic response defined as LVESV reduction ≥10% at 6 months after CRT-D implantation.
Clinical composite score CCS | 6 months
  CCS describing patients regardless of vital status at 6 months and includes both objective and subjective measures of clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Peraldo Neja, Principal Investigator — CORELAB Responsible; Cesare Aragno, Study Director — Kell s.r.l.
Locations (4):
- Italy (4):
  - S.Camillo de Lellis Hospital, Rieti
  - S.Eugenio Hospital, Rome
  - University Hospital Campus Bio-Medico, Rome
  - Fatebenefratelli Hospital, Rome